CLINICAL TRIAL: NCT04524299
Title: A Phase II,Randomized Controlled Clinical Trial of Staged Thoracic Radiotherapy Combined With Albumin Bound Paclitaxel and Nedaplatin Twice a Week for Locally Advanced NSCLC
Brief Title: Study of Radiotherapy Combined With Albumin Bound Paclitaxel and Nedaplatin for Locally Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1066
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; radiotherapy; albumin bound paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent chemotherapy Twice a Week (Experimental): During the period of radiotherapy, 30 mg / m2 albumin bound paclitaxel was intravenously infused twice a week for 0.5 hours, and nedaplatin 10 mg / m2 twice a week for 0.5 hours.
  Interventions: Radiation: chest radiation(IMRT); Drug: Concurrent chemotherapy twice a week
- Concurrent chemotherapy Once a Week (Active Comparator): During the same period of radiotherapy, albumin bound paclitaxel (50 mg / m2) was intravenously infused once a week for 0.5 hours; nedaplatin (25 mg / m2) was intravenously infused once a week for 0.5 hours.
  Interventions: Radiation: chest radiation(IMRT); Drug: Concurrent chemotherapy once a week

INTERVENTIONS:
Radiation: chest radiation(IMRT) — Patients will receive intensity modulated radiotherapy (IMRT) once a day, 5 days a week. The first stage: DT 3000 cGy / 6 FX; the second stage, DT 3500 cGy / 7 FX. Or: the first segment: DT 4000 cGy / 10 FX; the second segment DT 2400 cGy / 6 FX. The interval between two stages of radiotherapy was 4 weeks.
Drug: Concurrent chemotherapy twice a week — During the same period of radiotherapy, 30 mg / m2 albumin bound paclitaxel was intravenously infused twice a week for 0.5 hours, and nedaplatin 10 mg / m2 twice a week for 0.5 hours.
  1. When the radiotherapy dose was 3000 cGy / 6 FX + DT 3500 cGy / 7 FX, the infusion time was D1, D4, D8 of the first stage of radiotherapy; D1, D4, D8 of the second stage of radiotherapy.
  2. When the radiotherapy dose was 4000 cGy / 10 FX + DT 2400 cGy / 6 FX, the infusion time was D1, D4, D8, D11 of the first stage of radiotherapy; D1, D4, D8 of the second stage of radiotherapy
  Arms: Concurrent chemotherapy Twice a Week
Drug: Concurrent chemotherapy once a week — During the same period of radiotherapy, albumin bound paclitaxel (50 mg / m2) was intravenously infused once a week for 0.5 hours; nedaplatin (25 mg / m2) was intravenously infused once a week for 0.5 hours. The infusion time was D1, D8 of the first radiotherapy and D1, D8 of the second radiotherapy.
  Arms: Concurrent chemotherapy Once a Week

SUMMARY:
This phase II randomized study is to investigate the efficacy and toxicity of fractional thoracic radiotherapy combined with albumin bound paclitaxel and nedaplatin twice a week in the treatment of locally advanced non-small cell lung cancer compared with weekly chemotherapy.

DETAILED DESCRIPTION:
This phase II randomized study is to investigate the efficacy and toxicity of fractional thoracic radiotherapy combined with albumin bound paclitaxel and nedaplatin twice a week in the treatment of locally advanced non-small cell lung cancer compared with weekly chemotherapy.

Radiotherapy:

All patients will receive intensity modulated radiotherapy (IMRT) once a day, 5 days a week. The first stage: DT 3000 cGy / 6 FX; the second stage, DT 3500 cGy / 7 FX. Or: the first segment: DT 4000 cGy / 10 FX; the second segment DT 2400 cGy / 6 FX. The interval between two stages of radiotherapy was 4 weeks.

Concurrent chemotherapy:

The patients were randomly divided into two groups and received one of the following concurrent chemotherapy regimens:

Group A: during the same period of radiotherapy, 30 mg / m2 albumin bound paclitaxel was intravenously infused twice a week for 0.5 hours, and nedaplatin 10 mg / m2 twice a week for 0.5 hours.

1. When the radiotherapy dose was 3000 cGy / 6 FX + DT 3500 cGy / 7 FX, the infusion time was D1, D4, D8 of the first stage of radiotherapy; D1, D4, D8 of the second stage of radiotherapy.
2. When the radiotherapy dose was 4000 cGy / 10 FX + DT 2400 cGy / 6 FX, the infusion time was D1, D4, D8, D11 of the first stage radiotherapy, and D1, D4, D8 of the second stage radiotherapy.

Group B: during the same period of radiotherapy, albumin bound paclitaxel (50 mg / m2) was intravenously infused once a week for 0.5 hours; nedaplatin (25 mg / m2) was intravenously infused once a week for 0.5 hours. The infusion time was D1, D8 of the first radiotherapy and D1, D8 of the second radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer.
* There were measurable diseases according to recist1.1.
* Non operative stage III (AJCC / UICC eighth edition stage).
* When the lowest dose of radiotherapy was 60Gy, V20 > = 35% in both lungs.
* 18 years old or above, under 75 years old, regardless of gender.
* ECoG physical status score (see Annex 1) was 0-1.
* Initial treatment or chemotherapy.
* There was no previous chest radiotherapy, immunotherapy or biotherapy.
* Neutrophil absolute value ≥ 2000 cells / mm3, platelet ≥ 100000 cells / mm3
* Serum creatinine ≤ 1.25 times ULN or creatinine clearance rate ≥ 60 ml / min.
* Serum bilirubin ≤ 1.5 times ULN, AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN, alkaline phosphatase ≤ 5 times ULN.
* CB6 normal range.
* The patient and his family members agreed and signed the informed consent.

Exclusion Criteria:

* There were other malignant tumors in the past or during treatment, except for skin non melanoma or cervical carcinoma in situ.
* Any other disease or condition is contraindication to chemotherapy (e.g. active infection, within 6 months after myocardial infarction, symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia, immunosuppressive therapy).
* Pregnant or lactating women, women who did not undergo a pregnancy test (within 14 days before the first administration), and pregnant women.
* Bleeding tendency.
* Participants in other clinical trials within 30 days before the experiment.
* Drug addiction, long-term alcoholism and AIDS patients.
* There are uncontrollable seizures or loss of self-control due to mental illness.
* Patients with severe allergic history or specific constitution.
* The researchers consider that it is not suitable to participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
local control rate | 2 years
  To assess the efficacy of albumin bound paclitaxel twice a week in terms of local control rate for all patients

SECONDARY OUTCOMES:
Progression-free Survival | 2 Years
  To assess the efficacy of albumin bound paclitaxel twice a week compared with once a week in terms of progression-free survival
Overall Survival(OS) | 2 Years
  To assess the efficacy of albumin bound paclitaxel twice a week compared with once a week in terms of overall survival
Response Rate(RR) | 2 years
  To assess the efficacy of albumin bound paclitaxel twice a week compared with once a week in terms of response rate
Distant metastasis rate | 2 years
  To assess the efficacy of albumin bound paclitaxel twice a week compared with once a week in terms of distant metastasis rate
rate of grade 3-4 radiation esophagitis | 1 year
rate of grade 3-4 radiation pneumonitis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Prof., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Dillman RO, Seagren SL, Propert KJ, Guerra J, Eaton WL, Perry MC, Carey RW, Frei EF 3rd, Green MR. A randomized trial of induction chemotherapy plus high-dose radiation versus radiation alone in stage III non-small-cell lung cancer. N Engl J Med. 1990 Oct 4;323(14):940-5. doi: 10.1056/NEJM199010043231403. PMID 2169587
- [Background] Sause W, Kolesar P, Taylor S IV, Johnson D, Livingston R, Komaki R, Emami B, Curran W Jr, Byhardt R, Dar AR, Turrisi A 3rd. Final results of phase III trial in regionally advanced unresectable non-small cell lung cancer: Radiation Therapy Oncology Group, Eastern Cooperative Oncology Group, and Southwest Oncology Group. Chest. 2000 Feb;117(2):358-64. doi: 10.1378/chest.117.2.358. PMID 10669675
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Salama JK, Stinchcombe TE, Gu L, Wang X, Morano K, Bogart JA, Crawford JC, Socinski MA, Blackstock AW, Vokes EE; Cancer and Leukemia Group B. Pulmonary toxicity in Stage III non-small cell lung cancer patients treated with high-dose (74 Gy) 3-dimensional conformal thoracic radiotherapy and concurrent chemotherapy following induction chemotherapy: a secondary analysis of Cancer and Leukemia Group B (CALGB) trial 30105. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e269-74. doi: 10.1016/j.ijrobp.2011.01.056. Epub 2011 Apr 7. PMID 21477940
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Segawa Y, Kiura K, Takigawa N, Kamei H, Harita S, Hiraki S, Watanabe Y, Sugimoto K, Shibayama T, Yonei T, Ueoka H, Takemoto M, Kanazawa S, Takata I, Nogami N, Hotta K, Hiraki A, Tabata M, Matsuo K, Tanimoto M. Phase III trial comparing docetaxel and cisplatin combination chemotherapy with mitomycin, vindesine, and cisplatin combination chemotherapy with concurrent thoracic radiotherapy in locally advanced non-small-cell lung cancer: OLCSG 0007. J Clin Oncol. 2010 Jul 10;28(20):3299-306. doi: 10.1200/JCO.2009.24.7577. Epub 2010 Jun 7. PMID 20530281
- [Background] Desai N, Trieu V, Damascelli B, Soon-Shiong P. SPARC Expression Correlates with Tumor Response to Albumin-Bound Paclitaxel in Head and Neck Cancer Patients. Transl Oncol. 2009 May;2(2):59-64. doi: 10.1593/tlo.09109. PMID 19412420
- [Background] Desai N, Trieu V, Yao Z, Louie L, Ci S, Yang A, Tao C, De T, Beals B, Dykes D, Noker P, Yao R, Labao E, Hawkins M, Soon-Shiong P. Increased antitumor activity, intratumor paclitaxel concentrations, and endothelial cell transport of cremophor-free, albumin-bound paclitaxel, ABI-007, compared with cremophor-based paclitaxel. Clin Cancer Res. 2006 Feb 15;12(4):1317-24. doi: 10.1158/1078-0432.CCR-05-1634. PMID 16489089
- [Background] Green MR, Manikhas GM, Orlov S, Afanasyev B, Makhson AM, Bhar P, Hawkins MJ. Abraxane, a novel Cremophor-free, albumin-bound particle form of paclitaxel for the treatment of advanced non-small-cell lung cancer. Ann Oncol. 2006 Aug;17(8):1263-8. doi: 10.1093/annonc/mdl104. Epub 2006 Jun 1. PMID 16740598
- [Background] Rizvi NA, Riely GJ, Azzoli CG, Miller VA, Ng KK, Fiore J, Chia G, Brower M, Heelan R, Hawkins MJ, Kris MG. Phase I/II trial of weekly intravenous 130-nm albumin-bound paclitaxel as initial chemotherapy in patients with stage IV non-small-cell lung cancer. J Clin Oncol. 2008 Feb 1;26(4):639-43. doi: 10.1200/JCO.2007.10.8605. PMID 18235124
- [Background] Reynolds C, Barrera D, Jotte R, Spira AI, Weissman C, Boehm KA, Pritchard S, Asmar L. Phase II trial of nanoparticle albumin-bound paclitaxel, carboplatin, and bevacizumab in first-line patients with advanced nonsquamous non-small cell lung cancer. J Thorac Oncol. 2009 Dec;4(12):1537-43. doi: 10.1097/JTO.0b013e3181c0a2f4. PMID 19887966
- [Background] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591
- [Background] Socinski MA, Okamoto I, Hon JK, Hirsh V, Dakhil SR, Page RD, Orsini J, Yamamoto N, Zhang H, Renschler MF. Safety and efficacy analysis by histology of weekly nab-paclitaxel in combination with carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer. Ann Oncol. 2013 Sep;24(9):2390-6. doi: 10.1093/annonc/mdt235. Epub 2013 Jul 10. PMID 23842283
- [Background] Hasegawa T, Futamura Y, Horiba A, Yoshida T, Suzuki T, Kato T, Kaito D, Ohno Y, Iida T, Hayashi S, Sawa T. A phase II study of nab-paclitaxel plus carboplatin in combination with thoracic radiation in patients with locally advanced non-small-cell lung cancer. J Radiat Res. 2016 Jan;57(1):50-4. doi: 10.1093/jrr/rrv062. Epub 2015 Oct 5. PMID 26442970
- [Background] Lammers PE, Lu B, Horn L, Shyr Y, Keedy V. nab-Paclitaxel in Combination With Weekly Carboplatin With Concurrent Radiotherapy in Stage III Non-Small Cell Lung Cancer. Oncologist. 2015 May;20(5):491-2. doi: 10.1634/theoncologist.2015-0030. Epub 2015 Apr 6. PMID 25845992
- [Background] Kaira K, Tomizawa Y, Imai H, Sakurai R, Matsuura M, Yoshii A, Ochiai M, Kotake M, Ebara T, Saitoh JI, Sunaga N, Minato K, Saito R, Hisada T. Phase I study of nab-paclitaxel plus carboplatin and concurrent thoracic radiotherapy in patients with locally advanced non-small cell lung cancer. Cancer Chemother Pharmacol. 2017 Jan;79(1):165-171. doi: 10.1007/s00280-016-3217-1. Epub 2016 Dec 19. PMID 27995307
- [Background] Kawano Y, Sasaki T, Yamaguchi H, Hirano K, Horiike A, Satouchi M, Hosokawa S, Morinaga R, Komiya K, Inoue K, Fujita Y, Toyozawa R, Kimura T, Takahashi K, Nishikawa K, Kishimoto J, Nakanishi Y, Okamoto I. Phase I/II study of carboplatin plus nab-paclitaxel and concurrent radiotherapy for patients with locally advanced non-small cell lung cancer. Lung Cancer. 2018 Nov;125:136-141. doi: 10.1016/j.lungcan.2018.09.014. Epub 2018 Sep 18. PMID 30429011
- [Background] Gardner ER, Dahut WL, Scripture CD, Jones J, Aragon-Ching JB, Desai N, Hawkins MJ, Sparreboom A, Figg WD. Randomized crossover pharmacokinetic study of solvent-based paclitaxel and nab-paclitaxel. Clin Cancer Res. 2008 Jul 1;14(13):4200-5. doi: 10.1158/1078-0432.CCR-07-4592. PMID 18594000
- [Background] Wiedenmann N, Valdecanas D, Hunter N, Hyde S, Buchholz TA, Milas L, Mason KA. 130-nm albumin-bound paclitaxel enhances tumor radiocurability and therapeutic gain. Clin Cancer Res. 2007 Mar 15;13(6):1868-74. doi: 10.1158/1078-0432.CCR-06-2534. PMID 17363543